CLINICAL TRIAL: NCT06331637
Title: Postoperative and Functional Outcomes of Transanal Tran-section and Single-Stapled (TTSS) Ileal Pouch-Anal Anastomosis in Ulcerative Colitis Patients
Brief Title: Outcomes of Transanal Tran-section and Single-stapled (TTSS) Ileal Pouch-Anal Anastomosis
Acronym: TTSS-Pouch
Status: Not yet recruiting | Type: Observational
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Other Study IDs: 3782
Record Dates: First submitted 2024-03-19; First posted 2024-03-26 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Ulcerative Colitis
Keywords: Ileal Pouch-Anal Anastomosis; Intestinal Function
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Transanal Transection and Single-Stapled anastomosis (TTSS): Patients will undergo restorative proctectomy with Transanal Transection and Single-Stapled (TTSS) Ileal Pouch-Anal anastomosis (IPAA)
  Interventions: Procedure: Transanal Transection and Single-Stapled anastomosis (TTSS)
- Double-stapled anastomosis: Patients will undergo restorative proctectomy with double-stapled Ileal Pouch-Anal anastomosis (IPAA)
  Interventions: Procedure: Double-stapled anastomosis

INTERVENTIONS:
Procedure: Transanal Transection and Single-Stapled anastomosis (TTSS) — Restorative proctectomy with Transanal Transection and Single-Stapled (TTSS) Ileal Pouch-Anal Anastomosis (IPAA)
  Groups: Transanal Transection and Single-Stapled anastomosis (TTSS)
Procedure: Double-stapled anastomosis — Restorative proctectomy with Tdouble-stapled Ileal Pouch-Anal Anastomosis (IPAA)
  Groups: Double-stapled anastomosis

SUMMARY:
This study aims to compare the functional and surgical outcomes of Ulcerative Colitis (UC) patients undergoing Transanal Transection and Singl-Stapled (TTSS) versus Double-stapled Ileal Pouch-Anal Anastomosis (IPAA)

DETAILED DESCRIPTION:
Ileal Pouch-Anal Anastomosis (IPAAI in Ulcerative Colitis (UC) patients is usually performed by double-stapling technique after rectal transection with a linear stapler. Double-stapling is increasingly criticized for the uneven longer cuffs and potential weak points. The Transanal Transection and Single-Stapled (TTSS) approach may potentially overcome the limitations of double-stapling. A single-stapled anastomosis may be accomplished through a transanal rectal transection followed by bottom-up dissection (transanal-ileal pouch-anal anastomosis) or through an abdominal, rectal dissection and subsequent transanal transection and single-stapled anastomosis. TTSS-IPAA approach was shown to provide reduced rectal cuff length and reduced rate of urgency at six months after stoma closure. However, the retrospective and single-center features of these findings may prevent a robust conclusion about the superiority of TTSS-IPAA. The purpose of this study is to compare short-term and functional outcomes of double-stapling versus TTSS techniques for IPAA in UC patients in a prospective multicentric cohort study.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥ 18 years old) patients diagnosed with drug-refractory and/or steroid-dependent UC scheduled for elective restorative proctectomy.
* Patients scheduled for robotic or laparoscopic surgery

Exclusion Criteria:

* Planned open surgery.
* Concomitant colorectal cancer or dysplasia. Patients with an incidental intraoperative diagnosis of colorectal cancer will be withdrawn from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include adult patients diagnosed with drug-refractory and/or steroid-dependent Ulcerative Colitis (UC), scheduled for pouch surgery with double-stapled or Transanal Transection and Single-Stapled (TTSS) approach.
Sampling Method: Non-Probability Sample
Enrollment: 174 (Estimated)
Dates: Start 2024-07-31 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Pouch Function Score (PFS) | 6 months after surgery or stoma closure
  Median difference of the Pouch Function Score (PFS) [score ranging from 0 (no pouch symptoms) to 30 (severe pouch symptoms)] between the study cohorts

SECONDARY OUTCOMES:
Pouch Function Score (PFS) | 12 months after surgery or stoma closure
  Median difference of the Pouch Function Score (PFS) [score ranging from 0 (no pouch symptoms) to 30 (severe pouch symptoms)] between the study cohorts
Pouch Function Score (PFS) | 24 months after surgery or stoma closure
  Median difference of the Pouch Function Score (PFS) [score ranging from 0 (no pouch symptoms) to 30 (severe pouch symptoms)] between the study cohorts
Postoperative complications | 90 days after surgery
  Rate difference of postoperative complications, classified according to the Clavien-Dindo scale [ranging from 0 (no complications) to 5 (complications leading to death)] between the study cohorts
Anastomotic leak | 90 days after surgery
  Rate difference of anastotic leaks between the study cohorts
Patients fit for stoma closure | 12 months after surgery
  Proportion difference of patients fit for stoma closure in the study cohorts. Patients fit for stoma closure have already closed the stoma or have an intact anastomosis as demonstrated by a water contrast enema, Computed Tomography (CT) scan, endoscopic, or surgical revision
Healthcare costs | 12 months after surgery
  Median difference of healthcare costs (direct and indirect) between the study cohorts
Rectal cuff lenght | At surgery
  Median difference of rectal cuff lenght (in cm) between the study cohorts
Pouch complications | 24 months after surgery or stoma closure
  Incidence rate difference of pouch complications or defunction- defined as any condition affecting the pouch function or requiring the pouch breakdown, including acute or chronic pouchitis, cuffitis, Crohn's disease of the pouch, or any other inflammatory condition - between the study cohorts.

CONTACTS AND LOCATIONS:
Overall Officials: Antonino Spinelli, MD, PhD, Principal Investigator — Humanitas Research Hospital IRCCS, Rozzano-Milan
Locations (1):
- IRCCS Humanitas Research Hospital, Rozzano, MI, Italy

IPD SHARING:
Plan to Share IPD: No